CLINICAL TRIAL: NCT01942252
Title: COMPLICATIONS OF SECOND HAND SMOKING IN PEDIATRIC TONSILLECTOMY PATIENTS
Brief Title: COMPLICATIONS RELATED CARBOXYHEMOGLOBIN LEVELS IN SECOND HAND SMOKING PEDIATRIC TONSILLECTOMY PATIENTS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Onur Koyuncu, Asist.Prof.Dr., Mustafa Kemal University
Other Study IDs: 207; Onur Koyuncu (Registry Identifier: Onur Koyuncu)
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Secondhand Smoking
Keywords: Secondhand smoking, pain, postoperative complications
MeSH Terms: conditions — Pain; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study was to determine whether high carboxyhemoglobin level is a risk factor for postoperative adverse events in children exposured to carbon monoxide, especially enviromental tobacco smoke.

DETAILED DESCRIPTION:
Also we want to measure bleeding volume and compare it with the carboxyhemoglobin levels.

ELIGIBILITY:
Inclusion Criteria:

-Patients 1-12 years old scheduled for adenotonsillectomy; written informed consent.

Exclusion Criteria:

* Active smokers, history of prematurity, bleeding disorders, hemolysis, severe pulmonary disease, home oxygen use, and inpatient hospitalisation≥24 h.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Inclusion Criteria:
  -Patients 1-12 years old scheduled for adenotonsillectomy; written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Correlatin between carboxyhemoglobib levels of the second hand smoking children and postoperative complications and pain | Postoperative 24 hours

SECONDARY OUTCOMES:
Correlation between carboxyhemoglobin levels of the second hand smoking children and intraoperative bleeding volume | Intraoperative period
  Any relation between carboxyhemoglobin and bleeding?

OTHER OUTCOMES:
Correlation between carboxyhemoglobin levels and pain of the second hand smoking children | postoperative 24 hours
  Does second hand smoking affects pain?

CONTACTS AND LOCATIONS:
Overall Officials: ONUR KOYUNCU, ASSIST PROF, Study Director — Mustafa Kemal University
Locations (1):
- Mustafa Kemal University, Hatay, Turkey (Türkiye)

REFERENCES:
- [Result] Skolnick ET, Vomvolakis MA, Buck KA, Mannino SF, Sun LS. Exposure to environmental tobacco smoke and the risk of adverse respiratory events in children receiving general anesthesia. Anesthesiology. 1998 May;88(5):1144-53. doi: 10.1097/00000542-199805000-00003. PMID 9605672
- [Result] Koop CE. Adverse anesthesia events in children exposed to environmental tobacco smoke: exposure to environmental tobacco smoke and the risk of adverse respiratory events in children receiving general anesthesia. Anesthesiology. 1998 May;88(5):1141-2. doi: 10.1097/00000542-199805000-00001. No abstract available. PMID 9605670